CLINICAL TRIAL: NCT03367117
Title: Results of Peripheral Blood Stem Cells According to Stimulatory Molecule,: Zarzio Versus Granocytes
Acronym: ZAG
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ZAG
Record Dates: First submitted 2017-12-04; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-10

CONDITIONS: Hematology, Graft, Mobilization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigator therefore propose a retrospective mono-centric study, to compare the results obtained in patients with myeloma or lymphoma, mobilized with Zarzio® in order to obtain a graft, with the results obtained in our study. retrospective cohort of mobilization by Granocyte®.

DETAILED DESCRIPTION:
Autologous cell therapy remains the standard treatment in lymphomas (Hodgkin or non Hodgkin) and myelomas in the first line if they have bad prognostic factors or second-line cases of relapsed or relapsed patients. The essential condition for performing an autograft is the existence of a graft sufficient for this procedure. The European Society of Marrow Transplantation (EBMT) recommends to inject a minimum of 2 × 10 6 CD34 + cells / kg.

Although in terms of conventional products (Neupogen® and Granocyte®), the literature is very rich, there is no data on the use of biosimilars in this indication. A PUBMED search using the terms "peripheral blood stem cell harvest, OR Zarzio® biosimilars" did not produce any results.

Zarzio® has a tolerance and efficacy profile equivalent to "classical" products when used in post-chemotherapy, primary or secondary prophylaxis.

It therefore seems important to compare its efficacy and tolerance in mobilization situations for peripheral stem cell sampling.The Investigator therefore propose a retrospective mono-centric study, to compare the results obtained in patients with myeloma or lymphoma, mobilized with Zarzio® to obtain a graft, with the results obtained in our study. retrospective cohort of mobilization by Granocyte®.

ELIGIBILITY:
Inclusion Criteria:

* - Age supérieur to 8 year
* Recommandation of ABSCT

Exclusion Criteria:

* - No indication of ABSCT
* Age inférieur to 18 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lymphoma or myeloma patients for whom autologous stem cell tansplatation is a therapeutical option
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-01-23 (Actual)

PRIMARY OUTCOMES:
Stimulation by biosimilairs of Granulocyte - Colony stimulating factor ( G-CSF) | Two days
  Utilisation of bio similairs of GCSF for stimulation in view of obtaining an autologous graft